CLINICAL TRIAL: NCT06286189
Title: Effect of Trazodone on Obstructive Sleep Apnea Endotypes and Severity
Brief Title: Trazodone on OSA Endotypes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ludovico Messineo, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002760-t
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule 30 min before sleep
  Interventions: Drug: Placebo oral tablet
- Trazodone (Experimental): Trazodone capsule 30 min before sleep
  Interventions: Drug: Trazodone Hydrochloride

INTERVENTIONS:
Drug: Placebo oral tablet — Placebo capsule taken 30 min before sleep
  Arms: Placebo
Drug: Trazodone Hydrochloride — Trazodone 100 mg 30 min before sleep
  Arms: Trazodone

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. Some OSA patients with low arousal threshold wake up prematurely during an obstructive event and do not have time for spontaneous upper airway (UA) dilator muscle recruitment. As a consequence they are exposed to apnea and hypopnea cycling. In this protocol the investigators will test the effect of trazodone administered before sleep on OSA traits and OSA severity during sleep.

DETAILED DESCRIPTION:
Two overnight home sleep studies will be performed: a drug night and a placebo night. The patient will breath spontaneously (without CPAP) for both nights. On the study nights, subjects be instrumented with a full polygraphy for monitoring sleep, and respiratory events. Trazodone 100 mg will be given 30 min before lights out. At least four hours of sleep with high quality signal acquisition will be required for a study to be judged adequate. After the first overnight study is completed, there will be a one-week washout period prior to crossing over to the other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe OSA (AHI ≥ 15 events/hr)

Exclusion Criteria:

* All participants will be healthy and without major organ system disease that would preclude undergoing the physiological measurements.
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, acetazolamide, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Use of SNRIs/SSRIs.
* Conditions likely to affect OSA physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Sleep disordered breathing or respiratory disorders other than obstructive sleep apnea:
* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Hypersensitivity to the study drug (angioedema or urticaria)
* Contraindications to DAW2020
* Use of medications that lengthen QTc interval
* Hypokaliemia, hypomagnesemia, uncontrolled thyroid disease
* Severe claustrophobia.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of trazodone on arousal threshold (%eupnea) | 1 night
  Arousal threshold will be calculated non invasively from the home sleep test flow signal

SECONDARY OUTCOMES:
Effect of trazodone on apnea hypopnea index (events/h) | 1 night
  Apnea hypopnea index will be calculated from the home sleep test

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No